CLINICAL TRIAL: NCT06828835
Title: Testing a Strategy to Improve Diagnostic and Treatment Pathways for Children With Sleep-Disordered Breathing: the REPOSE Navigation Intervention
Brief Title: The REPOSE (Reach for Equity in Pediatric Sleep Evaluation) Navigation Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Phayvanh Pecha, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00138323; 1K23HL171952-01A1 (NIH)
Record Dates: First submitted 2025-02-05; First posted 2025-02-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Pediatrics; Sleep Disorders
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Wake Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reach for Equity in Pediatric Obstructive Sleep Evaluation (REPOSE) (Other): REPOSE is a theory-based patient navigation intervention to address multilevel barriers to timely diagnosis and treatment of obstructive sleep-disordered breathing.
  Interventions: Other: Reach for Equity in Pediatric Obstructive Sleep Evaluation (REPOSE)
- Usual Care (Other): The ordinary course of care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Reach for Equity in Pediatric Obstructive Sleep Evaluation (REPOSE) — The REPOSE intervention consists of a centralized patient navigator who (1) identifies and addresses dynamic individual barriers, (2) provides support for parent-child dyads, and (3) facilitates bidirectional SDB care coordination between clinical teams and parents to achieve evidence-based care. The goals of the REPOSE intervention are to systematically address barriers to care, develop parental self-efficacy to enhance healthcare utilization (e.g., receipt of recommended care and adherence to evidence-based care), and to improve symptom severity and quality of life.
  Arms: Reach for Equity in Pediatric Obstructive Sleep Evaluation (REPOSE)
Other: Usual Care — Usual care is defined by standard clinical care delivered without a protocolized intervention (e.g., the ordinary course of care).
  Arms: Usual Care

SUMMARY:
This research study aims to find out the effect of REPOSE, a patient navigation intervention, on the receipt of equitable care among children with a broad range of socioeconomic and rural/urban status with Sleep Disordered Breathing (SDB).

In the REPOSE intervention, a centralized patient navigator a) identifies and addresses dynamic individual barriers, b) provides resources and social support for parent-child dyads, and c) facilitates bidirectional SDB care coordination between clinical teams and parents to achieve evidence-based care.

This study will evaluate the effects of the REPOSE intervention on SDB care delivery and clinical process outcomes for children with a broad range of socioeconomic and rural/urban status by reducing barriers and increasing self-efficacy among parents.

DETAILED DESCRIPTION:
Sleep disordered breathing (SDB), defined as nocturnal respiratory disturbances ranging from snoring to severe obstructive sleep apnea, affects 12% children in the United States. The American Academy of Pediatrics recommends that all children be screened for snoring, and that those with symptoms or signs of SDB are further evaluated for medical treatment. Despite this recommendation, the rates for recognizing and screening SDB remain low. Black children are also 4-6 times more likely to have SDB but are less likely to undergo evaluation and to receive timely standard of care treatments to address their SDB. Untreated SDB is associated with significant health consequences including behavioral impairments, poor academic performance, and neurocognitive deficits. While evidence-based treatment is available, it is not accessible to all. Black children are 83% less likely than their White peers to attend consultations for SDB. A critical need exists for a theory-based intervention to reduce barriers to care for children with SDB.

Patient navigation is an evidence-based intervention that has been shown to improve screening, referral, and treatment in many health conditions and has high potential to be a culturally acceptable intervention to promote equity in the setting of racial disparities in SDB. Preliminary data informed the development of a novel, multilevel theory-based patient navigation intervention, Reach for Equity in Pediatric Obstructive Sleep Evaluation (REPOSE). In the REPOSE intervention, a centralized patient navigator a) identifies and addresses dynamic individual barriers, b) provides resources and social support for parent-child dyads, and c) facilitates bidirectional SDB care coordination between clinical teams and parents to achieve evidence-based care. In this hybrid type I effectiveness implementation study, the candidate will conduct a pilot randomized controlled trial (RCT) in which N=80 parent-child dyads will be randomized to REPOSE or usual care for SDB. The study team will examine the extent to which the REPOSE intervention improves rates of adherence to evidence-based guidelines among children with a broad range of socioeconomic and rural/urban status with SDB and changes in barrier resolution and self-efficacy among parents. In addition, barriers and facilitators to implementation will be evaluated as guided by the Consolidated Framework for Implementation Research (CFIR) with a focus on social determinants of health.

The findings of this randomized pilot trial will inform the design of a future fully powered RCT.

ELIGIBILITY:
Inclusion Criteria:

* Parents or caregivers (18 and older) of children who were referred by any primary care for SDB evaluation with sleep medicine or pediatric otolaryngology
* Patients 2.00 to 11.99 years old
* Parents with a working phone who are willing to participate in the study for a 12-month period after enrollment

Exclusion Criteria:

* Patients already established with sleep medicine or otolaryngology which would bias ease of completing specialty evaluation

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2026-02-03 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Completion of specialist evaluation | up to 12months
  Binary, evaluation of SDB by completion of specialist consultation (e.g., sleep medicine, otolaryngologist) per AAP guidelines.

SECONDARY OUTCOMES:
Time from referral to specialist consultation | 12months
  Time in days from referral order to specialist evaluation (sleep medicine or otolaryngology).
Completion of PSG | 12months
  Binary, PSG (if ordered) was completed within 90 days of the order.
Time to PSG | 12months
  Time in days from PSG order to completion.
Receipt of treatment | 12months
  Binary, treatment completion within 60 days.
Time to treatment | 12months
  Time in days from initial consultation or from PSG results to recommended treatment.
SDB symptom severity | 1-2 weeks following enrollment (T1), 12 months after enrollment (T3)
  Pediatric Sleep Questionnaire-Sleep-Related Breathing Disorder (PSQ-SRBD) Scale is a 22-item scale which measures symptoms of obstructive sleep apnea including snoring, observed apneas, difficulty breathing during sleep, daytime sleepiness, inattentive or hyperactive behavior, and other pediatric obstructive sleep apnea features. The responses are 0 "No" and 1 "Yes". The instrument is scored by averaging the response on non-missing items. A score greater than 0.33 corresponds to a high risk for a pediatric sleep-related breathing disorder.
Quality of life impact for obstructive sleep apnea in children | 1-2 weeks following enrollment (T1), 12 months after enrollment (T3)
  Sleep-specific quality of life; Obstructive Sleep Apnea (OSA-18) is an 18-item health-related quality of life survey to measure the quality- of-life impact for obstructive sleep apnea syndrome in children.
Barrier reduction | 1-2 weeks following enrollment (T1), 12months
  Proportion and types of barriers resolved.
Unresolved barriers | 12months
  Proportion of barriers unresolved by the navigator.
Self-efficacy | 1-2 weeks following enrollment (T1), 6 months after enrollment (T2)
  The NIH Toolbox Self-Efficacy Item Bank is a 10-item survey designed to assess the participant's belief in his or her capacity to manage problems and have control over meaningful events.

OTHER OUTCOMES:
Sociodemographic factors | Baseline (T0)
  Sex, age, race, ethnicity, SES, education, employment, income, distance to medical facility, rural/urban residence, and insurance status.
Clinical characteristics | Baseline (T0), 12months
  Comorbidities, body mass index (percentile), and PSG parameters.
Social Support | 1-2 weeks following enrollment (T1), 6 months after enrollment (T2)
  The Interpersonal Support Evaluation List (ISEL-12) is a 12-item measure of perceptions of social support with three subscale scores representing appraisal, belonging, and tangible social support.
REPOSE Accrual Rate | 12months
  REPOSE Accrual Rate is the proportion of eligible patients who enroll in REPOSE.
REPOSE Attrition Rate | 12months
  REPOSE Attrition Rate is the proportion of enrolled participants lost to follow-up over the study period.
Navigator Caseload | 12months
  Navigator Caseload is the number of simultaneous cases being navigated.
Navigator Time Allocation (Direct) | 12months
  Navigator Time Allocation (Direct) is the time (in minutes) that the navigator spends directly interacting with the patient to identify and address barriers to SDB care.
Navigator Time Allocation (Indirect) | 12months
  Navigator Time Allocation (Indirect) is the time (in minutes), that the navigator spends generating and enacting each Barrier Reduction Plan that is not directly interacting with the patient.
Study Questionnaire Completion Rate (Pre and Post) | 12months
  Study Questionnaire Completion Rate (Pre and Post) is the proportion of study questionnaires completed by enrolled study participants.
Feasibility of Intervention Measure (FIM) | 12 months after enrollment (T3)
  Feasibility of Intervention Measure (FIM) is a four-item tool that evaluates feasibility by measuring demonstrated content validity, reliability, structural validity, structural invariance, known-groups validity, and responsiveness to change.
Patient Satisfaction with Navigation | 12 months after enrollment (T3)
  Patient Satisfaction with Navigation (PSN-I questionnaire) is a validated, nine-item measure of the satisfaction with the interpersonal relationship with the patient navigator.
Acceptability of Intervention Measure (AIM) | 12 months after enrollment (T3)
  Acceptability of Intervention Measure (AIM) is a four-item tool that evaluates acceptability by measuring demonstrated content validity, reliability, structural validity, structural invariance, known-groups validity, and responsiveness to change.

CONTACTS AND LOCATIONS:
Overall Officials: Phayvanh Pecha, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States